CLINICAL TRIAL: NCT06686810
Title: Endoscopic Therapy in Patients With Primary Sclerosing Cholangitis: 30 Years of Experience
Brief Title: Endoscopy and Primary Sclerosing Cholangitis
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Tringali Andrea, MD, PhD, Assistant Professor of Surgery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3893
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: ERCP; Primary sclerosis cholangitis; biliary stricture; dominant biliary stricture; liver transplantation; balloon dilatation; cholangiocarcinoma
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing Endoscopic Retrograde CholangioPancreatyopgraphy for PSC: Patients undergoing Endoscopic Retrograde CholangioPancreatyopgraphy (ERCP) to dilate dominant biliary strictures related to Primary Sclerosing cholangitis (PSC)
  Interventions: Procedure: Endoscopic Retrogradade CholangioPancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic Retrogradade CholangioPancreatography (ERCP) — ERCP is an endoscopic therapeutic procedure to drain the bile ducts in case of stones or biliary strictures that can be treated by balloon dilatation or stents (plastic or metal) insertion

SUMMARY:
Primary Sclerosing Cholangitis (PSC) is a chronic, cholestatic, immune-mediated liver disease characterized by segmental inflammation, fibrosis and destruction of the intra and / or extrahepatic biliary tree.

Patients suffering from PSC can develop biliary strictures and symptoms (jaundice, itching, cholangitis) requiring endoscopic therapy by Endoscopic Retrograde Cholangiopancreatography (ERCP).

ERCP can play an important role in symptoms control, cholangiocarcinoma diagnosis.

PSC can lead to liver failure and subsequent need for liver transplantation, ERCP can therefore delay the time for liver transplantation.

With this work the investigators want to report our thirty years of experience in the endoscopic treatment of PSC.

DETAILED DESCRIPTION:
Population studies have provided an estimation of prevalence which is between 1-16 per 100,000 inhabitants. PSC occurs mainly in young adults between the ages of 25 and 45, although it can occur at any age.

There is a strong correlation between CSP and Chronic Inflammatory Bowel Diseases.

The etiology of PSC is not known, although its autoimmune origin is commonly accepted.

The onset of PSC is symptomatic in about 50% of cases and the presentation can range from non-specific symptoms (fatigue, itching, low-grade fever), to cholangitis or even to symptoms and signs of liver cirrhosis.

Of the imaging tests, MRCP , is the most accurate in the diagnosis of PSC and should be accompanied by periodic non-invasive evaluations of associated hepatic fibrosis.

There is currently no effective conservative treatment for the disease and therefore each approach is intended to alleviate cholestatic symptoms.

ERCP in the context of symptomatic treatment of the disease plays a fundamental role, because the endoscopic dilation of symptomatic dominant biliary stenosis is an effective, although temporary, therapeutic option in patients with PSC.

With this work we want to report our thirty years of experience in the endoscopic treatment of PSC.

The study will be conducted through the systematic retrospective analysis of the ERCP database carried out in the Digestive Endoscopy Unit of the Policlinico Gemelli IRCCS, Rome Italy and Department of Gastroenterology Hôpital Erasme, Cliniques universitaires de Bruxelles, Belgium, from 1983 to January 2020.

The following information will be sought:

* Patient age and sex.
* Indication to ERCP.
* Laboratory tests (cholestasis and cytolysis).
* Imaging tests performed (CT, MRCP).
* Diagnostic and therapeutic maneuvers carried out during ERCP (including sphincterotomy, dilations, brushing, stent placement or nasal-biliary tube) and possible failure.
* Anatomical description of the biliary tree during ERCP. The results of the treatment will be evaluated considering the time interval between one endoscopic treatment and the next as an index of symptomatic relapse and the report of outpatient visits carried out at the Hospital.

ERCP TECHNIQUE All procedures were performed by dedicated and experienced medical and nursing staff. Patients were placed in a prone or supine position for hilar and supra-hilar stenosis.

ERCP was performed under sedation with midazolam and fentanyl or directly under anesthesiology assistance.

Sphincterotomy and retrograde cholangiography with water-soluble contrast medium was performed in all patients. Selective antegrade cholangiography may have been performed in some patients with detailed MRCP.

The strictures were identified and treated by pneumatic dilatation (multiple, hilar and suprahilar stenoses) or by stent placement (single stenosis of the main biliary tract).

Brushing was performed, in accordance with current guidelines, when a new stenosis appeared or in case the stenosis presenting a morphology suspected for cholangiocarcinoma.

In case of stent placement, removal is scheduled within 15-90 days or when symptoms such as pain, jaundice, itching and cholangitis recur.

A nasal biliary drainage (NBD) placement at the end of the procedure to perform washing or collection of bile for cytology was performed, if needed, after pneumatic dilation procedures and / or in case of failure of stenting therapy.

STUDY DESIGN Observational, retrospective, non-profit study, which provides the collection in a dedicated database of clinical data deriving from the revision of the operating registers and the database of all ERCP performed in on PSC patients.

FOLLOW-UP Follow-up will be performed by telephone interview or preferably by clinical consultation.

The following data will be recoreded:

* Clinical conditions
* Presence of other morbid conditions such as chronic inflammatory bowel diseases and / or autoimmune diseases
* Latest lab / imaging data
* Administration of the Patient's Global Impression of Change (PGIC) scale questionnaire (15) aimed at assessing the quality of life after treatment

MANAGEMENT AND CONFIDENTIALITY OF THE COLLECTED DATA Patients candidates to the study, will receive an informed consent form for the processing of personal data and for participation in the study during office consultation. In the event that interview will be performed by telephone, verbal consent will be obtained.

These data will be collected in a specific database (processed by Excel ™, Microsoft Office 2020) anonymously, giving each patient only a progressive numerical code.

The owner of the processing of personal data will be the Digestive Endoscopy Unit of the Policlinico Gemelli IRCCS, Rome Italy and Department of Gastroenterology Hôpital Erasme, Cliniques universitaires de Bruxelles, Belgium and the person in charge is the principal investigator.

The data will be stored and analyzed anonymously and identified on the basis of the assigned numerical code. The data collected and processed will constitute the material for scientific publications, but also in this case the data will be reported anonymously.

The Head of the study and his collaborators will therefore have access to the data, who will in any case be bound by the obligation of confidentiality and data processing according to current regulations. The Ethics Committee and the Regulatory Authorities will have direct access to the medical documentation to verify the study procedures and / or the data to the extent required by current regulations.

STATISTICAL CONSIDERATIONS

Sample size: given the purely descriptive nature of the study, sample size can be hypothesized considering a sample of 90 patients, estimating, as reported in the literature, a success rate of 61% (55 patients) with a confidence interval of not less than 50% (95% CI, 50.% - 70%).

Statistical analysis: The sample will be described in its clinical characteristics (notes on clinical history, preoperative data and those concerning the procedure) and demographic through descriptive statistical techniques. Quantitative variables will be described through the following measures: minimum, maximum, range, mean and standard deviation. The qualitative variables will be described through tables of absolute and percentage frequencies.

The data obtained will be analyzed with MedCalc Statistical Software version 14.8.1 (MedCalc Software bvba, Ostend, Belgium; http://www.medcalc.org; 2014).

ETHICAL CONSIDERATIONS The protocol will be submitted to the Ethics Committee of the Digestive Endoscopy Unit of the Policlinico Gemelli IRCCS, Rome Italy and Department of Gastroenterology Hôpital Erasme, Cliniques universitaires de Bruxelles, Belgium for review and approval.

PUBLICATION POLICIES The preliminary and final results of the study will be collected and processed for presentation in national and international conferences and for the drafting of scientific papers for any publications. The authors of the scientific papers will be chosen according to the contribution made by them.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PSC and biliary tract stenosis with indication for endoscopic treatment.

Exclusion Criteria:

* Patients with unclear diagnosis of PSC.
* Patients ineligible for endoscopic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from primary sclerosis cholangitis and dominant biliary strictures with jaundice, cholangitis, suspicious of malignancy requiring endoscopic biliary drainage (balloon dilatation, scenting) and stricture sampling by ERCP
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of long-term endoscopic treatment | From Enrollment to the last follow-up, 3 years
  PSC can lead to liver failure and need for liver transplantation. Endoscopic therapy can have a positive impact to delay the need for liver transplantation

SECONDARY OUTCOMES:
Need for Endoscopic retreatment | From Enrollment to the last follow-up, 3 years
  Analyze rates of symptomatic disease recurrence (pain, jaundice, cholangitis, etc.) in terms of the need for retreatment after endoscopic therapy of PSC related biliary (pneumatic dilation in comparison with the placement of endoprostheses).
Occurrence of Cholangiocarcinoma | From Enrollment to the last follow-up, 3 years
  Analyze the incidence of cholangiocarcinoma in the course of PSC and the results of the brushing of the dominant biliary stenosis carried out in the course of ERCP
Adverse events | From Enrollment to the last follow-up, 3 years
  Incidence of adverse events related to endoscopic procedures (ERCP) (cholangitis, pancreatitis, bleeding, perforations)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tringali, MD, PhD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS Roma, Italy
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Endoscopia Digestiva, Roma, Italy